CLINICAL TRIAL: NCT06219408
Title: A Pilot Randomized Controlled Trial of CIH Stepped Care for Co-occurring Chronic Pain and PTSD
Brief Title: CIH Stepped Care for Co-occurring Chronic Pain and PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, David Reed, Assistant Professor: School of Medicine, Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00015530; R00AT012054 (NIH)
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Posttraumatic Stress Disorder
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: To mirror a future large-scale trial, the PI/biostatistician/randomizer will remain masked. An unmasked member of the research team will inform individuals to which group they are randomized and will be available to answer questions about assessments if needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIH Stepped Care (Experimental): CIH Stepped Care is a stepped approach to care delivered by a health coach (e.g., psychologist-in-training or clinical social worker) in-person or remotely (individual person sessions). It is a mindfulness-based and meaning-based stepped care approach for treating co-occurring chronic pain and PTSD that will begin with less intensive treatment (e.g., psychoeducation) and, based on patient response and preference, will be "stepped up" to more intensive treatment when appropriate.
  Interventions: Behavioral: CIH Stepped Care
- Treatment as Usual (No Intervention): Treatment as usual at the clinic

INTERVENTIONS:
Behavioral: CIH Stepped Care — CIH Stepped Care is a stepped approach to care delivered by a health coach (e.g., psychologist-in-training or clinical social worker) in-person or remotely (individual person sessions). It is a mindfulness-based and meaning-based stepped care approach for treating co-occurring chronic pain and PTSD that will begin with less intensive treatment (e.g., psychoeducation) and, based on patient response and preference, will be "stepped up" to more intensive treatment when appropriate.
  Arms: CIH Stepped Care

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, acceptability, appropriateness, and retention of patient participants of a CIH Stepped Care approach for co-occurring chronic pain and PTSD vs. treatment as usual in two primary care settings (one rural and one urban).

Researchers will compare CIH Stepped Care to treatment as usual.

Participants will complete assessments at baseline, 3-months, 6-months, and 9-months, and those in the CIH Stepped Care condition will participate in the intervention while also completed assessments every 2-weeks, which helps determine their treatment.

We hypothesize that, at 6-months, CIH Stepped Care will be feasible, acceptable, and appropriate (defined by an average of 4/5 on each measure) to patients and clinic employees and result in at least 70% of individuals be retained in each condition (n=21 per condition).

ELIGIBILITY:
Inclusion Criteria

In order to be eligible to participate in this study, clinic employees must meet all of the following criteria:

1. Aged 18 years or older
2. A clinic employee and/or trainee

In order to be eligible to participate in this study, patients must meet all of the following criteria:

1. Aged 18 years or older
2. English-speaking
3. A patient at the clinic from which recruitment occurs
4. Endorse chronic pain (defined as experiencing pain on more than half of the days of the past 3-months)
5. Endorse at least moderate pain severity and interference (defined as at least an average of 4 on the PEG)
6. Endorse at least 31 on the PCL-5, in combination with a Criterion A traumatic event. If we have difficulties in recruiting individuals who meet our PTSD diagnosis criteria, we will modify this criteria by removing the requirement of a Criterion A traumatic event, and require a destabilizing life event instead.

4.2 Exclusion Criteria

There are no exclusion criteria for clinic employees.

Patients who meet any of the following criteria will be excluded from participation in this study:

1. In current treatment for chronic pain and/or PTSD at their respective clinic
2. Past 2-week suicidal intention at screening
3. Severe cognitive impairment preventing individual from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure | 6-months
  Feasibility of intervention; 1-5; higher scores indicate greater feasibility
Acceptability of Intervention Measure | 6-months
  Acceptability of Intervention; 1-5; higher scores indicate greater acceptability
Appropriateness of Intervention Measure | 6-months
  Appropriateness of Intervention; 1-5; higher scores indicate greater appropriateness
Participant Retainment | 6-months
  Percentage of Participants Retained in Intervention Arm

SECONDARY OUTCOMES:
PTSD Diagnostic Scale for DSM-5 | Baseline, 3-, 6-, and 9-months
  PTSD symptoms; 0-80; higher scores indicate more severe PTSD symptoms
Patient Reported Outcome Measurement System - Pain Interference | Baseline, 3-, 6-, and 9-months
  Pain interference; 0-100; higher scores indicate worse pain interference

OTHER OUTCOMES:
PEG | Measurement-based care (every 2 weeks for those in CIH Stepped Care)
  Pain severity and interference; 0-10; higher scores indicate more pain severity and interference
Harvard's Flourishing Measure - Happiness and Life Satisfaction | Baseline, 3-, 6-, and 9-Months
  Happiness and Life Satisfaction; 0-10; higher scores indicate greater happiness and life satisfaction
Harvard's Flourishing Scale - Meaning and Purpose | Measurement-based care
  Meaning and Purpose (every 2 weeks for those in CIH Stepped Care); 0-10; higher scores indicate greater meaning and purpose
Emotion Regulation Questionnaire-Short Form | Baseline, 3-, 6-, and 9-months
  Cognitive re-appraisal; 3-21; higher scores indicate greater cognitive re-appraisal
Metacognitive Processes of Decentering Scale | Baseline, 3-, 6-, and 9-months
  Decentering; 0-10; higher scores indicate higher decentering
Meaning in Life Questionnaire | Baseline, 3-, 6-, and 9-months
  Meaning in Life; 1-7; higher scores indicate more meaning in life
Existential Phenomenological Questionnaire - Short Form | Baseline, 3-, 6-, and 9-months
  Existential Anxiety; 1-5; higher scores indicate more existential anxiety
Five Facet Mindfulness Questionnaire | Baseline, 3-, 6-, and 9-months
  Mindfulness; 24-120; higher scores indicate more mindfulness
Columbia-Suicide Severity Rating Scale - Self-Report | 3-, 6-, and 9-months
  Suicidality; 6 items; risk levels of high, moderate, low/no risk are determined
GAD-7 | Baseline, 3-, 6-, and 9-Months
  Anxiety; 0-21; higher scores indicate more severe anxiety symptoms
PHQ-9 | Baseline, 3-, 6-, and 9-Months
  Depression; 0-27; higher scores indicate more severe depression symptoms
PROMIS-Physical Health | Baseline, 3-, 6-, and 9-Months
  Physical Health; 0-100 T-scores; higher scores indicate greater physical health function
Working Alliance Inventory-Short Revised-Therapist | 3- and 6-months
  Therapeutic Alliance; 1-7; higher scores indicate greater working patient-provider therapeutic alliance
Reason for Dropout | 6-months
  1-item on why participant discontinued study
Fidelity of CIH Stepped Care | 6-months
  Treatment fidelity; percentage of items completed; greater percentage indicates higher fidelity
PTSD Checklist for DSM-5 | Measurement-based care (every 2 weeks for those in CIH Stepped Care)
  PTSD Symptoms; 0-80; higher scores indicate higher PTSD symptom severity
Adherence | 6-months
  Adherence (defined as completing over 50% of the measurement-based care assessments that occur every 2 weeks and completing participant-health coach measurement-based care contacts, where, for instance, treatment options would be discussed)
Medication use | Baseline, 3-, 6-, and 9-months
  Medication use (name, dose, and frequency)
Healthcare use | Baseline, 3-, 6-, and 9-months
  Healthcare use; frequency of different healthcare services used (e.g., primary care visits)
Treatment Change | Measurement-based care (every 2 weeks for those in CIH Stepped Care)
  1-item asking patients in the CIH Stepped Care condition whether they would like to change treatments
Working Alliance Inventory-Short Revised-Client | 3- and 6-months
  Therapeutic Alliance; 1-7; higher scores indicate greater working patient-provider therapeutic alliance

CONTACTS AND LOCATIONS:
Overall Officials: David Reed, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be de-identified and approved by the PI.
Time Frame: IPD and supporting information will be available after all data has been collected until data is destroyed.
Access Criteria: Researchers and others whose goal is to advance the science of improving care for those with chronic pain.